CLINICAL TRIAL: NCT03021707
Title: Early Feasibility Study of UV-Femtosecond Laser Assisted Lenticular Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RFO268-E001
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Refractive Error - Myopia Severe; Refractive Error - Myopia Simple

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- UV-FS laser (Experimental): WaveLight® Ultraviolet Femtosecond Laser System during UV-Femto, single session (one treatment per eye per participant)
  Interventions: Device: WaveLight® Ultraviolet Femtosecond (FS) Laser System; Procedure: Laser Assisted Lenticular Extraction

INTERVENTIONS:
Device: WaveLight® Ultraviolet Femtosecond (FS) Laser System — Utilizes ultraviolet (UV) light with a wavelength of 347 nanometers (nm) for refractive error correction
  Other Names: Model 1026; UV-FS laser
Procedure: Laser Assisted Lenticular Extraction — Used for refractive error correction
  Other Names: UV-Femto

SUMMARY:
The purpose of this study is to evaluate the initial safety of the UV-FS laser in humans.

ELIGIBILITY:
Inclusion Criteria:

* Photopic distance visual acuity worse than best corrected visual acuity (BCVA) 20/400 in the study eye;
* Myopia with manifest refraction spherical equivalent (MRSE) of - 1.50 diopter (D) or higher in the study eye;
* Able to comprehend and provide documented informed consent;
* Willing and able to comply with schedule for follow-up visits;
* Minimum required endothelial cell density (ECD) in study eye as outlined in the protocol;
* Presence of natural lens in study eye;
* A treatment simulation with spectacles or contact lenses on the study eye does not negatively impact participant's daily activities;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Pregnant or nursing;
* Acute or chronic disease or illness that would increase the operative risk or confound the outcomes of the study as clinically assessed by the Investigator;
* Active implanted device, including but not limited to, heart pacemaker or defibrillator, for which laser use may be a contraindication;
* Current use of medications with known ocular side effects;
* Predicted residual stromal bed thickness <300 micrometers (μm) in study eye
* Ocular conditions in the study eye;
* Previous ocular surgery in the study eye that resulted in corneal distortions within the treatment zone;
* Residual, recurrent or active ocular disease that may impact study outcomes;
* Previous or current diagnosis of dry eye;
* Known allergic reaction to medications expected to be used preoperatively, during laser refractive surgery, and for postoperative care;
* Pre-existing corneal opacities in study eye;
* Contact lens worn in study eye and not removed prior to study testing affected by wear per timeframe specified in the protocol;
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Presence of optical treatment zone corneal haze | Up to Month 6 (post-operative)
  Corneal haze will be assessed on a scale of 0 to 4, where 0 = clear or no haze can be seen, and 4 = opacity is visible without slit lamp, greatly obscures iris detail.
Mean change from screening in presence of disruption in the integrity of retinal layers in the macula | Screening, Up to Month 6 (post-operative)
  Retinal layer integrity will be assessed by a posterior segment ocular coherence tomography (OCT) scan of the study eye. Any disruption (change) in the retinal layers in the macula as compared to the screening scan will assess retinal integrity.
Mean percentage change in average endothelial cell density (ECD) from screening to each visit post procedure | Screening, Up to Month 6 (post-operative)
  Specular microscopy will be performed on the study eye and endothelial cell density will be recorded.
Mean percentage change in lens opacification from screening to each visit post procedure | Screening, Up to Month 6 (post-operative)
  A Scheimpflug scan will be performed to evaluate any opacification of the crystalline lens in the study eye and a Pentacam Nucleus Staging (PNS) grade from 0 to 5 will be assigned.
Mean percentage change in foveal thickness from screening to each visit post procedure | Screening, Up to Month 6 (post-operative)
  Foveal thickness will be assessed by a posterior segment OCT scan of the study eye.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, Surgical, Study Director — Alcon Research
Locations (4):
- United States (2):
  - Alcon Investigative Site, Sioux Falls, South Dakota
  - Alcon Investigative Site, Houston, Texas
- Alcon Investigative Site, Dublin, Ireland
- Alcon Investigative Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No